CLINICAL TRIAL: NCT06314659
Title: A Single-center, Randomized, Blind, Positive Control Phase III Clinical Trial to Evaluate Immunogenicity and Safety of Group A and C Meningococcal Polysaccharide Conjugate Vaccine in Volunteers Aged 3-5 Months
Brief Title: Immunogenicity and Safety of Group A and C Meningococcal Polysaccharide Conjugate Vaccine in Volunteers Aged 3-5 Months
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020020C
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Healthy Population
Keywords: Group A and C Meningococcal Polysaccharide Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic immunization (Experimental): Perform basic immunization with a program of 0, 1, and 2 months, booster vaccination with 1 dose at 18 months of age.
  Interventions: Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Zhifei Lvzhu); Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Walvax)
- Booster immunization (Active Comparator): Perform booster vaccination with 1 dose at 18 months of age.
  Interventions: Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Zhifei Lvzhu); Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Olymvax)

INTERVENTIONS:
Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Zhifei Lvzhu) — Performed primary immunization following a 0-1-2-month schedule at the aged from 3 to 5 months and booster immunization at 18 months of age.
Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Walvax) — Performed primary immunization following a 0-1-2-month schedule at the aged from 3 to 5 months.
  Arms: Basic immunization
Biological: Group A and C Meningococcal Polysaccharide Conjugate Vaccine (producted by Olymvax) — Performed booster immunization at 18 months of age.
  Arms: Booster immunization

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Group A and C Meningococcal Polysaccharide Conjugate Vaccine in healthy volunteers aged from 3 to 5 months old.

DETAILED DESCRIPTION:
This is a Phase III, single center, randomized, blind, positive control clinical trial conducted in Guangxi Province, China. The purpose of this study is to evaluate the immunogenicity and safety of Group A and C Meningococcal Polysaccharide Conjugate Vaccine in healthy volunteers aged from 3 to 5 months old. A total of 630 subjects were included and randomly assigned to the experimental group and control group in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

For primary immunization stage

* Subjects aged 3-5 months;
* Subjects should be full-term (37-42 weeks of gestation) and their birth weight should meet the requirements (2500g ≤ body weight ≤ 4000g);
* Axillary body temperature ≤ 37.0 ℃;
* The guardian signs the informed consent form;
* The guardian and his family agree to comply with the requirements of the clinical trial protocol;
* Subjects who have not been vaccinated with meningococcal group A and C conjugate vaccine;
* Subjects who had no history of other live vaccines within 14 days before vaccination and no history of other inactivated vaccines within 7 days;

For booster immunization and immune persistence stage

* Infants in the experimental group who have completed primary immunization in this clinical trial and reach the age of 18 months;
* Infants and young children who have completed primary or booster immunization in this clinical trial;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

Exclusion Criteria:

For primary immunization stage

* Test-tube baby who is suffering from perianal abscess, severe eczema or pathological jaundice;
* History of severe allergic reactions requiring medical intervention (such as swelling of mouth and throat, dyspnea, hypotension or shock);
* A clearly diagnosed history of thrombocytopenia or other coagulation disorders that may cause contraindications to intramuscular injection;
* History of severe abnormal labor and delivery, asphyxia rescue, congenital malformation, serious developmental disorder, serious genetic defect, serious malnutrition or serious chronic disease;
* Suffering from serious cardiovascular diseases (pulmonary heart disease, pulmonary edema), serious liver and kidney diseases, and diabetes with complications;
* Has been diagnosed as infectious diseases, such as tuberculosis, viral hepatitis or their parents infected with human immunodeficiency virus (HIV);
* History or family history of encephalopathy, epilepsy, convulsions or seizures, and other progressive neurological diseases;
* Suffering from acute illness or in the acute phase of chronic illness, or using antipyretic, analgesic, and antiallergic drugs (such as acetaminophen, ibuprofen, aspirin, etc.) three days before vaccination;
* Long term treatment with immunosuppressants, such as long-term (continuous for more than 2 weeks) use of glucocorticoids (such as prednisone or inhaled steroids (budesonide, fluticasone) and similar drugs);
* History of using immunoglobulins and / or any blood products (except hepatitis B immunoglobulin) within 3 months before enrollment;
* Plan to participate or be participating in any other drug clinical research;
* Plan to move out of the local area before the end of the study or leave for a long time during the scheduled study visit period;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

For booster immunization and immune persistence stage

* Has been vaccinated with any meningococcal vaccine after primary immunization and before blood collection of booster immunization;
* Has been vaccinated with any meningococcal vaccine after booster immunization and before blood collection of immune persistence;
* Has been known or suspected to have immunological defects since participating in this clinical trial, including being treated with immunosuppressants (such as chemotherapy, corticosteroids, antimetabolics, cytotoxic drugs, etc.) and HIV infection;
* History of using immunoglobulins and / or any blood products within 3 months before booster immunization;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 630 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of antibody positivity conversion rate of serogroup A | 30 day after primary immunization
  The proportion of people with pre-immunization antibody titer against serogroup A meningococcus <1:8 who achieve an antibody titer ≥1:8 after immunization.
Analysis of antibody positivity conversion rate of serogroup C | 30 day after primary immunization
  The proportion of people with pre-immunization antibody titer against serogroup C meningococcus <1:8 who achieve an antibody titer ≥1:8 after immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi, China